CLINICAL TRIAL: NCT03317743
Title: Open-label, Phase I Clinical Trial to Identify Optimal Dose and Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics and the Anti-cancer Efficacy of NOV140101(IDX-1197HCl) in Patients With Advanced Solid Tumors
Brief Title: Study to Assess the Safety & Tolerability of NOV140101(IDX-1197) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idience Co., Ltd. (Industry)
Collaborators: IlDong Pharmaceutical Co Ltd (Industry); National OncoVenture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV140101-101/ID-VDP-101
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumors
Keywords: 1197; IDX-1197; venadaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOV140101 (IDX-1197) (Experimental)
  Interventions: Drug: NOV140101 (IDX-1197)

INTERVENTIONS:
Drug: NOV140101 (IDX-1197) — The dose levels will be escalated following a 3+3 dose escalation scheme.

SUMMARY:
the purpose of this open-label, dose escalation-dose expansion, Phase 1 clinical trial is to evaluate the safety, pharmacokinetics and anti-tumor activity and determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of NOV140101 (IDX-1197).

DETAILED DESCRIPTION:
This is an open-label, Phase 1 dose escalation study of NOV140101 (IDX-1197) to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and the anti-tumor efficacy of IDX-1197 in patients with advanced solid tumors after failure of standard of care. DLTs will be assessed as the primary endpoint in this trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 year old patients with histologically or cytologically confirmed metastatic or unresectable advanced solid tumors
* Life expectancy ≥12 weeks
* Women of childbearing potential must have a negative pregnancy test outcome
* ECOG performance status ≤2
* Lesions measured by tumor markers or CT/MRI and evaluable according to RECIST v1.1
* Patient must have adequate organ function as indicated by the following laboratory values independent of transfusion within 2 weeks:

  1. ANC ≥ 1,500/mm³
  2. Platelet count ≥ 100,000/mm³
  3. Hemoglobin ≥ 9.0g/dL
  4. Serum creatinine ≤ 1.5×ULN
  5. Total bilirubin ≤ 1.5×ULN
  6. AST, ALT ≤ 3×ULN (≤ 5×ULN for patients with liver metastasis or liver cell cancer)
  7. PT and aPTT ≤ 1.5×ULN
  8. UPC < 1.0 g/g (one re-test is allowed if positive (≥ 1))
* Patients must provide written informed consent to voluntary participation in this study.

Exclusion Criteria:

* History of hypersensitivity reactions to any of the components of the investigational product or other drugs of the same class
* New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled hypertension (systolic/diastolic blood pressure >140/90mmHg), or other clinically significant cardiovascular abnormalities in the opinion of the investigator
* Uncontrolled cardiac arrhythmia
* Acute coronary syndrome (unstable angina pectoris or myocardial infarction) within the past 6 months
* Major electrocardiogram (ECG) abnormalities in the opinion of the investigator
* Severe infection or severe traumatism
* Pneumonia or respiratory symptoms, such as dyspnea, cough, and fever, requiring treatment and other conditions likely to be accompanied by hypoxemia
* History of drug or alcohol abuse within the past 3 months
* Symptomatic or uncontrolled central nervous system (CNS) metastasis
* Less than 4 weeks have elapsed since a major surgery and 2 weeks have elapsed since a minor surgery
* Radiotherapy, hormone therapy, or chemotherapy within 2 weeks prior to baseline from which toxicities not recovered to ≤grade 1
* >4 weeks of persistent Grade 3 (NCI-CTCAE v4.03) hematologic toxicities from prior anticancer treatment
* History of myelodysplastic syndrome (MDS) or pre-treatment cytogenetic test results indicative of the risk of MDS or acute myelocytic leukemia
* Ongoing or anticipated treatment with antiplatelet drugs (aspirin, clopidogrel, etc.) or anticoagulant drugs (warfarin, heparin, etc.) during the study
* Requiring continuous treatment with systemic NSAIDs or systemic corticosteroids
* Ongoing or past treatment with immunosuppressants within 14 days prior to the first dose of study treatment, except for intranasal, inhaled, topical, or locally injected (e.g., intraarticular injection) steroids
* History of serious gastrointestinal bleedings within 12 weeks prior to screening or presence of diseases that may affect oral drug absorption (e.g., malabsorption syndrome, active peptic ulcer)
* History of human immunodeficiency virus infection or active hepatitis B or C infection or ongoing uncontrolled chronic infectious disease
* Pregnant or lactating women or patients planning to become pregnant during the study
* Participation in another clinical trial within 30 days prior to screening
* Individual considered ineligible for this study for other reasons, in the opinion of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-10-13 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-21)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- [Derived] Kim SB, Bae KS, Lee JL, Lee WS, Ock CY, Lee MJ, Bang J, Hong MJ, Roh EJ, Ha KS, Lim JH, Kim YM. First-In-Human Dose Finding Study of Venadaparib (IDX-1197), a Potent and Selective PARP Inhibitor, in Patients With Advanced Solid Tumors. Cancer Med. 2025 Feb;14(4):e70576. doi: 10.1002/cam4.70576. PMID 39945311